CLINICAL TRIAL: NCT05266365
Title: Investigation of the Efficacy of Video-Based Exercise Programs in Degenerative Meniscus Tears
Brief Title: The Video-Based Exercise Programs in Degenerative Meniscus Tears
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 107
Record Dates: First submitted 2022-02-28; First posted 2022-03-04 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Degenerative Disease; Meniscus Tear; Knee Pain Swelling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Video-based exercise (VBE) group (Experimental): Each subject in the video-based exercise group (only video-based intervention) will receive a treatment protocol consisting of stretching, strengthening, and functional exercises for the knee and hip.
  Interventions: Other: The video-based exercise (VBE)
- The standard exercise (SE) group (Active Comparator): Each subject in the standard exercise group (only clinic-based intervention) will receive a treatment protocol consisting of stretching, strengthening, and functional exercises for the knee and hip.
  Interventions: Other: The standard exercise (SE)
- The hybrid exercise (HE) group (Experimental): Each subject in the hybrid exercise group (video-based and clinical-based interventions) will receive a treatment protocol consisting of stretching, strengthening, and functional exercises for the knee and hip.
  Interventions: Other: The hybrid exercise (HE)

INTERVENTIONS:
Other: The video-based exercise (VBE) — An 8-week exercise program will be implemented as part of the conservative treatment for degenerative meniscal tears. The physiotherapist will prepare an instructional video that provides a detailed explanation and demonstration of each exercise. Patients will watch this video at home and perform the exercises according to the video instructions.
  Arms: The Video-based exercise (VBE) group
Other: The standard exercise (SE) — An 8-week exercise program used in conservative treatment of degenerative meniscus tears will be performed.
  An exercise program will be performed at the clinic.
  Arms: The standard exercise (SE) group
Other: The hybrid exercise (HE) — An 8-week exercise program will be implemented as part of the conservative treatment for degenerative meniscal tears using a hybrid telerehabilitation model. For the home-based component, the physiotherapist will prepare an instructional video that includes a detailed description and demonstration of each exercise. Patients will watch this video at home and perform the prescribed exercises by following the instructions provided in the video. In addition to the home program, patients will also participate in supervised exercise sessions conducted in the clinical setting.
  Arms: The hybrid exercise (HE) group

SUMMARY:
This randomized controlled trial aims to investigate the efficacy of the video-based exercise programs in patients with degenerative meniscus tears.

DETAILED DESCRIPTION:
To investigate the efficacy of video-based exercise programs, voluntary patients with degenerative meniscus tears aged 40-65 years will be randomly assigned to three groups: the hybrid exercise group (HEG), the video-based exercise (VBE) group, and the standard exercise (SE) group. Interventions will be delivered over 16 sessions (twice a week for 8 weeks). The patients will be assessed at baseline and at the end of the 8-week intervention. Pain during activity, at rest, and at night will be assessed using the Visual Analog Scale (VAS). Active range of motion will be evaluated using a digital goniometer. Isometric muscle strength will be measured with a handheld dynamometer. The Knee Injury and Osteoarthritis Outcome Score (KOOS) will evaluate functional status and symptoms. The Western Ontario Meniscal Evaluation Tool (WOMET) will assess health-related quality of life. Adherence to the exercise program and the Global Rating of Change Scale will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 40 and 65 years
* Having the degenerative meniscus tear in at least one knee
* Having body mass index in the range of 18-30 kg/m2
* Feeling the pain that lasts for at least 2 months
* Having grade 1 or grade 2 degenerative meniscal tear diagnosed by an orthopedic specialist according to the MRI results
* Having the activity level is between 1 and 5 according to the Tegner Activity Scale
* Having access to the internet via a computer or smartphone
* Having the ability to read and write Turkish

Exclusion Criteria:

* Having undergone arthroscopic partial meniscectomy surgery due to degenerative meniscal tear
* Participating in a physiotherapy program for degenerative meniscal tear in the last 12 weeks
* Have received steroid injections in the last 6 months
* Accompanying conditions such as injury to the surrounding ligaments, congenital anomaly in the affected knee, coxarthrosis and spinal stenosis
* Presence of any systemic disorder that may affect assessment parameters
* Failure to cooperate with assessments
* Any vision or hearing problem that would prevent them from adapting to the assessment

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline
  Short-term and long-term symptoms and function will be assessed with the Knee injury and Osteoarthritis Outcome Score (KOOS) that is developed as an extension of the WOMAC Osteoarthritis Index. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | At the end of 8-week intervention
  Short-term and long-term symptoms and function will be assessed with the Knee injury and Osteoarthritis Outcome Score (KOOS) that is developed as an extension of the WOMAC Osteoarthritis Index. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Visual Analogue Scale (VAS) | Baseline
  Pain intensity will be measured using the visual analogue scale (VAS). The participants will be asked to indicate their perceived pain at rest, during activity and at night on the 10 cm line between no pain and terrible pain. The score will be determined by measuring the distance on 10 cm line using a ruler. The higher scores indicate an higher level of pain.
Visual Analogue Scale (VAS) | After 8-week intervention
  Pain intensity will be measured using the visual analogue scale (VAS). The participants will be asked to indicate their perceived pain at rest, during activity and at night on the 10 cm line between no pain and terrible pain. The score will be determined by measuring the distance on 10 cm line using a ruler. The higher scores indicate an higher level of pain.
Active Range of Motion | Baseline
  Active knee range of motion including flexion and extension will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a digital goniometer.
Active Range of Motion | At the end of 8-week intervention
  Active knee range of motion including flexion and extension will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a digital goniometer.
Muscle Strength | Baseline
  Isometric muscle strength will be measured with a handheld dynamometer for knee flexors and extensors. The process will be repeated three times in each direction, with the average value recorded.
Muscle Strength | At the end of the 8-week intervention
  Isometric muscle strength will be measured with a handheld dynamometer for knee flexors and extensors. The process will be repeated three times in each direction, with the average value recorded.
Western Ontario Meniscal Evaluation Tool (WOMET) | Baseline
  The health-related quality of life related to degenerative meniscal tear will be used with the WOMET, which is a disease-specific tool designed to evaluate health-related quality of life in patients with meniscal pathology. The WOMET contains sixteen items addressing three domains: nine items addressing physical symptoms; four items addressing disabilities due to sports, recreation, work, and lifestyle; and three items addressing emotions. The best and least symptomatic score is 0, and the highest and most symptomatic score possible is 1600.
Western Ontario Meniscal Evaluation Tool (WOMET) | At the end of the 8-week intervention
  The health-related quality of life related to degenerative meniscal tear will be used with the WOMET, which is a disease-specific tool designed to evaluate health-related quality of life in patients with meniscal pathology. The WOMET contains sixteen items addressing three domains: nine items addressing physical symptoms; four items addressing disabilities due to sports, recreation, work, and lifestyle; and three items addressing emotions. The best and least symptomatic score is 0, and the highest and most symptomatic score possible is 1600.

OTHER OUTCOMES:
Global Rating of Change | At the end of 8-week intervention
  The Global Rating of Change is a single-item self-report measure used to assess the participant's perceived overall change following the intervention. At the end of the 8-week intervention, participants will be asked to rate how their current condition compares to their condition before the treatment.
Adherence to Exercise Programs | Throughout the 8-week intervention period
  Adherence to the video-based exercise program will be monitored using daily participant-completed exercise logs and verified by weekly video submissions demonstrating the performance of selected exercises. The physiotherapist will directly monitor adherence to the clinic-based exercise program.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, PhD, PT, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No